CLINICAL TRIAL: NCT05088733
Title: Yang Yin Fu Zheng Jie Du Therapy in HBV Related Hepatocellular Carcinoma Induced Anemia
Brief Title: Yang Yin Fu Zheng Jie Du Therapy in HBV Related Hepatocellular Carcinoma Induced Anemia (YYFZJDTIHBVRHCIA)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Zhiyun Yang, Archiater, Professor, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJDHYZY
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yang Yin Fu Zheng Jie Du therapy (Experimental)
  Interventions: Drug: Yang Yin Fu Zheng Jie Du therapy; Other: Routine medical care
- Routine medical care (Placebo Comparator)
  Interventions: Other: Routine medical care

INTERVENTIONS:
Drug: Yang Yin Fu Zheng Jie Du therapy — Yang Yin Fu Zheng Jie Du is a Chinese herbal compound.
  Arms: Yang Yin Fu Zheng Jie Du therapy
Other: Routine medical care — Routine medical care

SUMMARY:
Clinical research of Yang Yin Fu Zheng Jie Du therapy in HBV related hepatocellular carcinoma induced anemia. The purpose of this study is to observe the efficacy of routine medical care combined with Yang Yin Fu Zheng Jie Du therapy for patients belong to HBV-HCC induced anemia.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of hepatocellular carcinoma
* Patients who tested positive for hepatitis B surface antigen (HBsAg) for >6 months
* Meet the criteria of anemia
* Ages Eligible for Study: ≤75 years old;
* Informed consent from the patient.

Exclusion Criteria:

* Patients with upper gastrointestinal bleeding within 3 months before enrollment;
* History of blood transfusion within 3 months before enrollment;
* Patient with other chronic hepatopathy, such as AIH, NAFLD, ALD;
* Serious problem of heart, lung, or kidney with severe dysfunction;
* Pregnant or child breast feeding women;
* Mental or cognitive disorders;
* Participating in other drug trials;
* Who are allergic to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 1 year

SECONDARY OUTCOMES:
Objective response rate | 1 year
quality of life (QOL) questionnaire | 1 year
  The questionnaire includes appetite, sleep, fatigue, pain, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiyun Yang, Beijing, Beijing Municipality, China